CLINICAL TRIAL: NCT05699954
Title: Assessment of the Blink (First) Impression Regarding the Presence of Cancer Within Colorectal Polyps
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0488
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Polyp; Colorectal Cancer; Colono
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Presence of Blink impression features for cancer in colorectal polyps — 1. 20 LNPCPs will be collected from the UZ Ghent database (all LNPCPs, ICF present).
  2. A survey will be made where participant endoscopist will be informed about the study. They will here be asked for electronic consent.
  3. The survey asks for demographics of the participant endosopists (experience, country where they work).
  4. The last part of the survey is where the 20 images of the LNPCPs are shown. After evere image 4 questions are asked. Is this a colorectal polyp? (Yes/No)
     * Is your Blink (first) Impression that this polyp contains cancer? (Yes/No)
     * If "yes", why do you think that? (Free comment box)
     * What treatment would you recommend for this polyp? (piecemeal endoscopic mucosal resection/endoscopic submucosal disection/surgery)
  5. Study will be closed after 2 weeks.
  6. Data analysis

SUMMARY:
Colorectal cancer (CRC) is a leading cause of death in the Western world. It can be effectively prevented by removal of pre-malignant polyps during colonoscopy. Large (≥20mm) non-pedunculated colorectal polyps (LNPCPs) represent 2-3% of colorectal polyps and require special attention prior to treatment. If submucosal invasive cancer (SMI) is suspected, careful decision making is required to exclude features which unacceptably increase the risk of lymph node metastases and render local treatment (endoscopic) non-curative. Such patients require a multi-disciplinary approach and consideration of surgery +/- systemic therapy.

Unfortunately, current classification systems are complex, require extensive training and technology not available in the majority of non-tertiary hospitals. They are therefore underused leading to incorrect decision making and negative patient outcomes (e.g. piecemeal resection without the chance of endoscopic cure or unnecessary further procedures in referral centres with resultant surgery anyway or surgery for benign disease).

Studies from the field of psychology show that humans are often capable of making correct decision based on their Blink (first) impression. It is also suggested that this Blink impression is based on experience and training. This might suggest that experienced or specialist endoscopist are better at diagnosing SMI within colorectal polyp at Blink impression.

The investigators hypothesize that by training the Blink impression, endoscopist of varying experience are able to detect cancer within LNPCPs. This can be proven by assessing the Blink impression of endoscopist of varying experience regarding the presence of SMI within LNPCPs.

Increasing the accuracy of the determination of SMI within colon polyps would directly translate into improvements in patient care and outcome.

For example, if SMI is present and is not suspected, patients may undergo unnecessary endoscopic procedures for an LNPCP which will eventually require surgery anyway (inconvenience, delayed correct treatment). If the incorrect technique is performed in the context of superficial SMI, adequate assessment of complete excision or extent and type of SMI may not be possible and a patient who would otherwise have been cured may require surgery anyway (under-treatment, below standard of care outcome, delay to treatment). Conversely, if SMI is suspected in its absence patients may undergo unnecessary surgery, increased healthcare spends and mortality (over-treatment, unnecessary risk). If the presence of SMI could be accurately determined in real-time using endoscopic imaging, delays to treatment, over-treatment and the associated morbidity for patients could be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists of varying abilities and grades (participant endoscopist) that consents electronically
* Patients with LNPCPs who signed the ICF of UZ Ghent Hospital for the anonymous use images of their polyp taken during colonoscopy

Exclusion Criteria:

* Endoscopist does not consent to inclusion (participant endoscopist)
* Image of inadequate quality as per opinion of the principal investigator
* Patient does not consent to data collection for the study (participant patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Endoscopists of varying experience (trainees, consultants, expert endoscopists, interventional endoscopists.
  * Patients with LNPCPs
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of endoscopic assessment as to the risk of SMI within LNPCPs. | Through study completion, Study is open for 2 weeks
  The accuracy of endoscopic assessment as to the risk of SMI within LNPCPs, using the Blink (first) impression when analysing images of LNPCPs.

SECONDARY OUTCOMES:
Identifying the parameters of LNPCPs that prompt endoscopist to have a positive Blink impression for the presence of SMI. | Through study completion, Study is open for 2 weeks
  Identifying the parameters of LNPCPs that prompt endoscopist to have a positive Blink impression for the presence of SMI.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No